CLINICAL TRIAL: NCT05998369
Title: Empowered Relief for Youth: A Feasibility Study of a Pain Management Class for Youth With Pain
Brief Title: Empowered Relief for Youth
Acronym: ER-Y
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Laura E Simons, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68451
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Musculoskeletal Pain; Fibromyalgia; Neuropathic Pain; Complex Regional Pain Syndromes; Abdominal Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain; Fibromyalgia; Neuralgia; Complex Regional Pain Syndromes; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empowered Relief for Youth (Experimental): Empowered Relief for Youth is a single-session pain management class focused on pain science education and teaching self-regulatory skills for pain management based on the evidence-based adult ER class.
  Interventions: Behavioral: Empowered Relief for Youth

INTERVENTIONS:
Behavioral: Empowered Relief for Youth — The Empowered Relief for Youth is a 90-minute class that provides pain science education, as well as cognitive, emotional, and physiologic self-regulation skills for youth with chronic pain. Youth will also develop a personalized plan to use the acquired skills daily. Participants will receive an audio file (Relaxation Response) post-class. The class provides patients rapid access to actionable skills for symptom management and pain relief.

SUMMARY:
The purpose of this pilot study is to examine the feasibility and preliminary efficacy of Empowered Relief for Youth with chronic pain (ER-Y). ER-Y is a single-session pain management class for youth focused on pain science education and teaching self-regulatory skills for pain management based on the evidence-based adult ER class. Feasibility and acceptability of ER-Y will be assessed post-class. Preliminary efficacy will be assessed by administering surveys at baseline, 4-weeks, 8-weeks, and 12-weeks post class.

DETAILED DESCRIPTION:
The current proposed, single-arm, uncontrolled pilot study will determine a) feasibility of ER-Y in youth with chronic pain, b) patients' perceptions and satisfaction of the ER-Y class and c) preliminary efficacy to inform the design of a subsequent randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 10 years old to 18 years
* Diagnosis of Chronic Pain
* English speaking

Exclusion Criteria:

* Significant psychosocial complexity (e.g., severe depression/ anxiety, unable to tolerate a group setting)
* non-English Speaking

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Treatment Expectancy Credibility (TEC-C) | Immediately post class
  The TEC-C assess treatment expectations and credibility with standardized sum scores from using a numeric rating scale (score 0 = "not at all" to 10 = "very much") with a higher score indicating high expectations.
Program Feedback Scale | Immediately post class
  The Program Feedback Scale assesses participants agreement to seven statements indicating their perceived acceptability and feasibility based on a scale (score 0 = "really disagree" to 4 = "really agree") with a higher score indicating positive feedback and two open ended questions.

SECONDARY OUTCOMES:
PROMIS Pain Interference | Pre class, 4 weeks, 8 weeks, and 12 weeks post class
  The PROMIS Pain Interference form assesses to what level pain hinders their engagement in several activities using a ranked scale (score 0 = "never" to 4 = "almost always") with a higher score indicating great pain interference.
Patient Global Impression of Change (PGIC) | 4 weeks, 8 weeks, and 12 weeks post class
  The Pain Global Impression of Change survey asks participants to rank how their overall pain has changed since the start of study using a ranked scale (score 0 = "very much improved" to 6 = "very much worse") with higher scores indicating greater severity to their pain.
Pain Catastrophizing Scale (PCS) | Pre class, 4 weeks, 8 weeks, and 12 weeks post class
  The Pain Catastrophizing Scale -Child Version (PCS-C, Crombez et al., 2003) assesses negative cognitions associated with pain. The PCS-C is comprised of 13-items rated on a 5-point Likert scale (score 0= "not at all true" to 4 "very true"). A total score (0-52) is obtained by summing all items. Higher scores indicate higher levels of catastrophic thinking.

OTHER OUTCOMES:
Child Pain Self-Efficacy Scale (PSES-C) | Pre class, 4 weeks, 8 weeks, and 12 weeks post class
  The Child Pain Self- Efficacy Scale assesses the participants self-efficacy with regard to normal functioning when in pain based on a ranked scale (score 1 = "very sure" to 5 = "very unsure") with higher scores indicating enhanced uncertainty.
PROMIS Anxiety | Pre class, 4 weeks, 8 weeks, and 12 weeks post class
  The PROMIS anxiety study assesses fear, fear, misery, hyperarousal, and somatic symptoms related to arousal within the past seven days. Each item is scored on a 1-5 rating scale (score 1 = "never" to 5 = "almost always") with higher scores indicating greater experience to anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Simons, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States